CLINICAL TRIAL: NCT02808702
Title: Brain Correlates of Self-Focused Processing as a Biomarker of Treatment Response
Brief Title: Brain Correlates of Self-Focused Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angela Fang, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1K23MH109593-01 (NIH)
Record Dates: First submitted 2016-06-08; First posted 2016-06-22 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Social Phobia; Body Dysmorphic Disorder
Keywords: Attention; Cognitive behavioral therapy; Neuroimaging
MeSH Terms: conditions — Phobia, Social; Body Dysmorphic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive-behavioral therapy (Experimental): Twelve weekly sessions of individual cognitive-behavioral therapy
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Twelve weekly sessions of individual cognitive-behavioral therapy

SUMMARY:
The purpose of this study is to determine whether neuroimaging-based markers of maladaptive self-focused processing are better predictors of treatment response to cognitive-behavioral therapy than behavioral markers.

DETAILED DESCRIPTION:
First, the investigators propose to identify the neural correlates of self-focused processing. The investigators will assess baseline resting state connectivity within the default network, as well as regional brain activation using a well-validated event-related fMRI task that manipulates self-focused processing in patients with body dysmorphic and socially anxious symptoms, compared to healthy controls. This clinical sample was selected because such patients display heightened self-focused attention, and sampling individuals across these symptom dimensions will ensure greater variability on this dimension of maladaptive self-focused processing. Second, the investigators will examine the neural correlates of self-focused processing as a predictor of treatment response. Neuroimaging data will be acquired from patients with body dysmorphic and socially anxious symptoms during two scan sessions, before and after 12 weeks of individual cognitive behavioral therapy, and compared with healthy controls scanned twice at a 12 week interval. Finally, the investigators will compare the prediction of treatment response between neural measures and behavioral measures of self-focused processing. The investigators will assess the behavioral correlates of self-focused processing using a self-reference effect paradigm, and assess their relation to treatment response. If the investigators hypotheses are borne out, the investigators will have new targets for treatment, a method to identify promising candidates for treatment, and sensitive surrogate markers of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18-45
* For patients: treatment-seeking individuals presenting with at least moderate levels of social anxiety/body dysmorphic symptoms, and a score of at least 1 SD above the mean on the public self-consciousness scale of the Self-Consciousness Scale- Revised
* For healthy controls only: no current or lifetime history of psychiatric disorders, and score of below 1 SD of mean on the SCS-R
* Right-handed, as determined by the Handedness Inventory
* Fluent in English, and willing to provide informed consent

Exclusion Criteria:

* Positive MR screen
* History of head injury, neurological disorder, or neurosurgical procedure
* Active suicidal or homicidal ideation
* Current or past manic/hypomanic episode or psychotic symptoms
* Active alcohol and substance dependence (as assessed by the SCID-5-RV
* Current use of psychotropic medications, except antidepressants taken at a stable dose for 2 weeks, to maximize generalizability of sample
* Current CBT and/or formal mindfulness/meditation training
* History of more than 10 sessions of CBT and formal mindfulness/meditation training

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline clinical symptoms at 12 weeks | Baseline and 12 weeks from baseline
  Evidence of symptom improvement as determined by clinician-administered assessment of body dysmorphic and socially anxious symptoms
Neural activation in the default mode network | Baseline and 12 weeks later
  Difference in regional brain activation in the default mode network in the Self vs. Other contrast (specifically in the medial prefrontal cortex, temporoparietal junction, posterior cingulate) during fMRI activation paradigm
Resting state functional connectivity within the default mode network | Baseline and 12 weeks later
  Functional connectivity within the default mode network during resting state scan
Response latencies during Self vs. Other conditions | Baseline and 12 weeks later
  Difference in average response latencies (in ms) during Self and Other conditions of a self-referential processing task

SECONDARY OUTCOMES:
Word valence during Self vs. Other conditions | Baseline and 12 weeks later
  Number of positive and negative words endorsed during Self and Other task conditions
Structural connectivity within the default mode network | Baseline and 12 weeks later
  White matter connectivity within the default mode network during DTI scan

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fang, Ph.D., Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fang A, Baran B, Feusner JD, Phan KL, Beatty CC, Crane J, Jacoby RJ, Manoach DS, Wilhelm S. Self-focused brain predictors of cognitive behavioral therapy response in a transdiagnostic sample. J Psychiatr Res. 2024 Mar;171:108-115. doi: 10.1016/j.jpsychires.2024.01.018. Epub 2024 Jan 16. PMID 38266332
- [Derived] Fang A, Baran B, Feusner JD, Phan KL, Beatty CC, Crane J, Jacoby RJ, Manoach DS, Wilhelm S. Self-Focused Brain Predictors of Cognitive Behavioral Therapy Response in a Transdiagnostic Sample. medRxiv [Preprint]. 2023 Sep 2:2023.08.30.23294878. doi: 10.1101/2023.08.30.23294878. PMID 37693433
- [Derived] Fang A, Baran B, Beatty CC, Mosley J, Feusner JD, Phan KL, Wilhelm S, Manoach DS. Maladaptive self-focused attention and default mode network connectivity: a transdiagnostic investigation across social anxiety and body dysmorphic disorders. Soc Cogn Affect Neurosci. 2022 Jul 2;17(7):645-654. doi: 10.1093/scan/nsab130. PMID 34875086